CLINICAL TRIAL: NCT06957496
Title: Phleum Pratense and Dactylis Glomerata Allergen Extracts. Determination of the in Vivo Histamine Equivalent Prick Test Units
Brief Title: Phleum Pratense and Dactylis Glomerata Allergen Extracts Standardization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inmunotek S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: G110-STD-071
Record Dates: First submitted 2024-09-16; First posted 2025-05-04 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Allergy Pollen; Allergic Reaction; Allergic Skin Reaction
Keywords: Allergy
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Phase II trial, open-label, prospective, non-randomized, without a control group of subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phleum pratense extract + Dactylis glomerata extract + positive control + negative control (Experimental): There is only one treatment arm. In each subject, one drop of each of the three concentrations of both allergenic extracts, along with the positive (histamine) and negative (saline solution) controls, will be applied to each subject.
  Phleum pratense: 100, 10 and 1 µg/mL Dactylis glomerata: 100, 10 and 1 µg/mL
  Interventions: Other: Allergenic extracts

INTERVENTIONS:
Other: Allergenic extracts — In each subject, a drop of each of the 3 concentrations of the allergenic extract, in addition to the positive control (histamine) and the negative control, will be applied. The application will be duplicated on the subject's anterior forearm, with a distance of approximately 4 cm between each application to avoid overlapping reactions and false-positives results.
  Other Names: Phleum pratense and Dactylis glomerata extracts

SUMMARY:
The primary objective is to assess the concentration of each allergen extract (Phleum pratense and Dactylis glomerata) that induces a wheal size equivalent to that produced by a 10 mg/mL histamine dihydrochloride solution. The standardization procedure is carried out according to the Aas Method as specified in the guideline developed by the Nordic Council on Medicines

DETAILED DESCRIPTION:
The trial will consist of a single visit, in which the following procedures will be carried out:

* Demographic data (age, race, and gender).
* Medical history: Time of onset of allergic rhinitis, rhinoconjunctivitis, allergic asthma and sensitizations (positive skin prick test) to allergens other than Phleum pratense and Dactylis glomerata.
* Inclusion/exclusion criteria.
* Physical examination (Cardiovascular, pulmonary, neurobiological, gastrointestinal, dermatological, other body systems and height, weight).
* Pregnancy test. Women of childbearing age will undergo a urine pregnancy test.
* Performance of prick-tests (3 concentrations of Phleum pratense and Dactylis glomerata allergenic extracts, positive control and negative control).
* Collection of blood sample (20 mL) from the subjects to create a pool of sera for the "in vitro" standardization of the allergenic extracts. Each serum sample will be stored in a tube labeled with the subject number and frozen. These serum samples will remain in the freezer until the end of the study. When the study is completed, they will be transported to the laboratory, where all sera will be pooled. This "pool" of sera will be used to perform the complementary in vitro tests necessary to standardize and characterize this extract and produce its corresponding IHRP (In-house reference preparation), as indicated by the Royal Spanish Pharmacopoeia and the European Pharmacopoeia. In addition, it will be used in the in vitro analyses necessary for the standardization of new batches of this allergenic extract. Once the pool has been formed, the tubes containing the original serum samples are destroyed.
* Assesment of adverse events. The trial will also include a follow-up call 72 hours after the prick tests are performed to monitor possible adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have signed and dated informed consent form.
* Female or male aged 18 to 64 years, both included.
* Subjects must reside in a geographical area where allergic problems caused by Phleum pratense and Dactylis glomerata are relevant.
* Positive medical history of inhalant allergy (rhinitis and/or rhinoconjunctivitis and/or asthma) to Phleum pratense and Dactylis glomerata.
* A positive prick-test (mean wheal diameter ≥ 3 mm) with extracts of the same allergens and/or presence of specific IgE against complete extract or any molecular component to the allergenic sources.
* The area of the wheal obtained with 10 mg/mL histamine dihydrochloride should be ≥ 7 mm², which corresponds to a mean wheal diameter ≥ 3 mm.
* The area of the wheal obtained with negative control should be < 7 mm², which corresponds to a mean wheal diameter < 3 mm.
* Women of childbearing age (i.e following menarche and until postmenopause, defined as no menses for 12 months without an alternative medical cause, or non-subject to permanent sterilization methods, such as hysterectomy, bilateral salpingectomy, and bilateral oophorectomy) must present a negative urine pregnancy test at the time of enrollment in the trial, as well as a confirmed menstrual period.
* Women of childbearing age must commit to using a highly effective and adequate contraception method during the trial and up to 72 hours after the end of treatment with the investigational medicinal product. Such methods include combined (estrogen and progestogen containing) hormonal; contraception associated with inhibition of ovulation (oral, intravaginal, or transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable), intrauterine device, intrauterine hormone-releasing system, male condom, diaphragm used with spermicide, bilateral tubal occlusion, vasectomized partner or sexual abstinence.

Exclusion Criteria:

* Subjects outside the age range.
* Subjects who have previously received immunotherapy within the last 5 years for the treatment of asthma or allergic rhinoconjunctivitis induced by allergens that may interfere with the extracts of Phleum pratense and Dactylis glomerata.
* Subjects with significant symptoms of rhinoconjunctivitis and/or bronchial asthma in whom discontinuation of systemic antihistamine treatment is contraindicated.
* Subjects who have previously exhibited a severe adverse reaction during diagnostic skin prick tests.
* Subjects on treatment with ß-blockers.
* Use of drugs that could interfere with skin prick test reactions (e.g., antihistamines) (See Section 5.2).
* Clinically unstable subjects (acute asthma, febrile, etc.).
* Subjects with active urticaria lesions, severe active dermographism, severe atopic dermatitis, sunburn, eczema, psoriasis lesions in the area where the prick test is performed (risk of false positives).
* Subjects with active herpes simplex viral infection, or herpes varicella zoster in the area where the prick test is performed.
* Subjects with any pathology in which the administration of adrenaline is contraindicated (hyperthyroidism, hypertension, heart disease, etc.).
* States in which the subject is unable to offer cooperation and severe psychiatric disorders.
* Pregnant or potentially pregnant women and breastfeeding women.
* Subjects with known phenol allergy.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-01-16 (Actual)

PRIMARY OUTCOMES:
Skin induced wheal measurement | 15 minutes after allergen introduction
  Measure of the area (mm^2) of the induced wheal on the skin upon applying each of the 3 concentrations of each allergenic extract (Phleum pratense and Dactylis glomerata), as well as those induced by positive (histamine) and negative controls, through the prick test.

SECONDARY OUTCOMES:
Adverse events registration | Through study completion, an average of 6 months
  Registration of any adverse events that occurred during the course of the trial
Adverse reactions registration | Through study completion, an average of 6 months
  Registration and documentation of any adverse reaction that occurred during the course of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Ojeda, Principal Investigator — Clínica de Asma y Alergia Dres. Ojeda
Locations (1):
- Clínica de Asma y Alergia Dres. Ojeda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No